CLINICAL TRIAL: NCT02488031
Title: Dysmetria in Motor Function in SCA: Mechanisms and Rehabilitation
Brief Title: Functional and Structural Imaging and Motor Control in Spinocerebellar Ataxia
Acronym: SCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201500202-N; R21NS094946 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Spinocerebellar Ataxia
Keywords: SCA, dysmetria
MeSH Terms: conditions — Spinocerebellar Ataxias; Heart Arrest; Cerebellar Ataxia | interventions — Weights and Measures; Stroop Test; Walking; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Error-reduction (Experimental): The participants in the error-reduction group will participate in a 4-week home-based training intervention during the month between their pre- and post-test visits. During pre- and post- training visits, Cooperative Ataxia Rating Scale (ICARS) and the Scale for the Assessment and Rating of Ataxia (SARA), Purdue Pegboard, Brief Test of Attention, 6-minute Walk, Hand Grip Dynamometer, Physical Performance Function, Digit Span, SARA, Montreal Cognitive Assessment, Beck Depression Inventory 2nd Ed, Stroop and biomechanical gait analysis tests will be administered. Also biomechanical assessments of dysmetria and neurophysiological assessment of brain activity will be conducted to evaluate the impact of the training on SCA individuals.
  Interventions: Behavioral: Error-reduction; Behavioral: International Cooperative Ataxia Rating Scale; Behavioral: Scale for the Assessment and Rating of Ataxia; Behavioral: Beck Depression Inventory, 2nd Ed; Behavioral: Stroop; Behavioral: Purdue Pegboard; Behavioral: Brief Test of Attention; Behavioral: 6-minute Walk; Behavioral: Hand Grip Dynamometer; Behavioral: Montreal Cognitive Assessment; Behavioral: Physical Performance Function; Behavioral: Biomechanical Assessments of Dysmetria; Behavioral: Neurophysiological assessment of brain activity; Behavioral: Biomechanical gait analysis
- Best Medical Management (Experimental): The participants in the best medical management group will undergo identical testing sessions (two visits one month apart) as those in the error-reducing group but will not receive the 4-week error reducing intervention. They will be administered the International Cooperative Ataxia Rating Scale (ICARS) and the Scale for the Assessment and Rating of Ataxia (SARA) assessments and the following tests: Purdue Pegboard, Brief Test of Attention, 6-minute Walk, Hand Grip Dynamometer, Physical Performance Function, Digit Span, SARA, Montreal Cognitive Assessment, Beck Depression Inventory 2nd Ed, Stroop and biomechanical gait. Biomechanical assessments of dysmetria and neurophysiological assessment of brain activity will be conducted at both visits.
  Interventions: Behavioral: International Cooperative Ataxia Rating Scale; Behavioral: Scale for the Assessment and Rating of Ataxia; Behavioral: Beck Depression Inventory, 2nd Ed; Behavioral: Stroop; Behavioral: Purdue Pegboard; Behavioral: Brief Test of Attention; Behavioral: 6-minute Walk; Behavioral: Hand Grip Dynamometer; Behavioral: Montreal Cognitive Assessment; Behavioral: Physical Performance Function; Behavioral: Biomechanical Assessments of Dysmetria; Behavioral: Neurophysiological assessment of brain activity; Behavioral: Biomechanical gait analysis

INTERVENTIONS:
Behavioral: Error-reduction — During this time participants will use a novel, custom designed computer interface to perform goal-directed movements with each leg in a 3D virtual environment designed to emphasize accurate movements. Leg movement will be detected using the LeapMotion sensor and we will quantify time endpoint errors by comparing the timing of the foot trajectory and the required time to target.
  The error-reduction intervention will be a 4-week home-based program. Each participant will train 4 days a week for approximately 1 hours per day. Within a week, the task difficulty will increase by changing the presentation of the targets to be more unpredictable and by increasing movement speed.
  Arms: Error-reduction
Behavioral: International Cooperative Ataxia Rating Scale — The ICARS is an assessment of the ataxia severity. The ICARS score is the total sum of the sub scores on specific movements and ranges from 0 to 100, with a score of 100 being indicative of the most severely affected outcome.
Behavioral: Scale for the Assessment and Rating of Ataxia — The SARA is an assessment of the ataxia severity. The SARA score is the total sum of the sub scores on specific movements and ranges from 0 to 100, with a score of 100 being indicative of the most severely affected outcome.
  Other Names: SARA
Behavioral: Beck Depression Inventory, 2nd Ed — This is a 21 question self-report inventory for measuring severity of depression.
Behavioral: Stroop — This test measures selective attention and cognitive flexibility through reading aloud of color names or color of the print.
Behavioral: Purdue Pegboard — This test consists of a series of timed hand coordination and dexterity tasks.
Behavioral: Brief Test of Attention — A cognitive test assessing focus and attention.
Behavioral: 6-minute Walk — This test consists on a timed 6-minute walk test to evaluate how much distance is covered.
Behavioral: Hand Grip Dynamometer — This tests measures hand grip strength.
Behavioral: Montreal Cognitive Assessment — This test is used to assess cognitive abilities.
Behavioral: Physical Performance Function — This test consists of a series of physical activities used to evaluate speed, coordination, and ease of movement.
Behavioral: Biomechanical Assessments of Dysmetria — Dysmetria will be assessed using a custom-made goal-directed movement protocol where participant perform unloaded limb movement tasks and attempt to reach a space-time target. During these task muscle activity is monitored using Electromyography (EMG) recording.
Behavioral: Neurophysiological assessment of brain activity — Neurophysiology will be assessed by monitoring brain activity using Task-based fMRI and motor unit pool activity using a specialized EMG system.
Behavioral: Biomechanical gait analysis — Participants will wear APDM's wireless sensors on the hands, legs, trunk and forehead and walk overground a distance of 7 m for 2 minutes. APDM quantifies 80 common biomechanical outcomes of gait (e.g. stride length variability).

SUMMARY:
The purpose of this research study is to investigate how the brain and motor behavior changes both in individuals with spinocerebellar ataxia and healthy individuals, and to assess whether a therapeutic intervention reduces levels of uncoordinated movement and improves motor function in spinocerebellar ataxia (SCA).

DETAILED DESCRIPTION:
Thirty individuals who have been diagnosed with either Spinocerebellar Ataxia - 1 (SCA1), Spinocerebellar Ataxia - 3 (SCA3), or Spinocerebellar Ataxia - 6 (SCA6) will be recruited for this study. Participants will be randomly assigned to a best medical management (BMM / control) group and an error-reduction group. All participants will visit the lab twice for testing one month apart. Participants in the control group will not train between the pre- and post-test time.

The error-reduction intervention will be a 4-week home-based program. Investigators will use a novel, custom designed computer interface. Participants will perform goal-directed movements with each leg to targets in a 3D virtual environment designed to emphasize accurate movements. The goal-directed leg movements (similar to leg press) will be performed seated and require hip, knee, and ankle joint control. Leg movement will be detected using the LeapMotion sensor (Leap Motion Inc. San Francisco, CA), a device that supports hand, and finger / tool motions as input, similar to a mouse, but requiring no contact. Spatial endpoint errors will be quantified in 3D space by comparing the endpoint location of the foot trajectory (extending from the big toe) and the virtual location of the target. Time endpoint errors will be quantified by comparing the timing of the foot trajectory and the required time to target.

The length of the intervention will be 4 weeks. Each participant will train 4 days a week for ~1 hour per day. Within a week the task difficulty will increase by changing the presentation of the target from a predictable to an unpredictable location, by increasing movement speed requirements and by changing target size. Targets will be made predictable by identifying them prior to the cue for movement onset (target turning green). Specifically, there will be a flashing dotted line around the target prior to the target turning green. Targets will be made unpredictable by not providing any indication of the target location prior to the target turning green. Movement speed will be quantified from the voluntary movement onset of the leg (no reaction time) to the movement end.The movement speed requirements will be increased within a week and participants will learn to execute faster movements from the feedback after each trial. The size of the target will be progressively reduced during the 4 weeks.

All individuals in the study will receive a pre- and post-test assessment using the International Cooperative Ataxia Rating Scale (ICARS) and the Scale for the Assessment and Rating of Ataxia (SARA). The individual sections of the ICARS (e.g. Kinetic section) and SARA will be quantified.

In addition, leg dysmetria will be quantified using a custom-made goal-directed movement protocol. Specifically, participants will perform unloaded ankle dorsiflexion movements and attempt to reach a space-time target. The primary outcomes will be position and time errors.

Biomechanics of overground walking in SCA will be monitored using the APDM mobility lab (APDM, Inc. Mobility Lab, Oregon, USA). Participants will wear APDM's wireless sensors on the hands, legs, trunk and forehead and walk overground a distance of 7 meters for 2 minutes. APDM quantifies 80 common biomechanical outcomes of gait (e.g. stride length variability).

The neurophysiology of SCA will be quantified with functional Magnetic Resonance Imaging (fMRI) and motor unit pool activity. Brain activity will be quantified with task-based fMRI using a 32-channel head coil. During fMRI force tasks, ankle dorsiflexion will be measured from the most affected lower limb using customized fiber optic sensors, as has been done in the past. Real-time feedback of force performance will be provided to the subject. During the rest blocks, subjects will fixate on a stationary target but do not produce force. During task blocks, subjects will complete 2 second pulse-hold contractions to 15% maximum voluntary contraction(MVC) of ankle dorsiflexion followed by 1 second of rest. There will be 10 pulses per block. The knee will be supported by a pillow to flex the knee so that the forces applied by the ankle do not cause head movement.

ELIGIBILITY:
Inclusion Criteria:

* DNA diagnosis of SCA1, SCA3, or SCA6
* phenotype consistent with the DNA diagnosis
* ability to walk 7 meters
* the age of 21-85 years
* capable of providing informed consent and complying with the trial procedures

Exclusion Criteria:

* Known recessive, X-linked or mitochondrial ataxias or any other type of ataxia
* Concomitant disorder(s) that affect ataxia measures used in this study
* Cognitive status on the Montreal Cognitive Assessment < 24
* Patients who have any type of implanted electrical device (such as a cardiac pacemaker or a neurostimulator), or a certain type of metallic clip in their body (i.e., an aneurysm clip in the brain), and are not eligible for participation in the MRI portion of the study
* Individuals who are claustrophobic
* Women who are or might be pregnant and nursing mothers
* Individuals with psychiatric disorders or dementia, along with other neurological and orthopedic problems that impair hand movements and walking

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03; Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Change in the Location of the Movement Endpoint Relative to the Target in the Motor Task | Change from Baseline to 1 month
  Assessment of the subject's ability to stay on target during the motor task. The task is a goal-directed movement that aims to match a spatial target in a specific time(time target).

SECONDARY OUTCOMES:
International Cooperative Ataxia Rating Scale(ICARS) Assessment | Change from Baseline to 1 month
  The ICARS is an assessment of the ataxia severity. The ICARS score is the total sum of the sub scores on specific movements and ranges from 0 to 100, with a score of 100 being indicative of the most severely affected outcome.
Change in Motor Unit Discharge Rate Variability | Change from Baseline to 1 month
  Amount of motor unit activity occurring during the Electromyography(EMG) task. Lower amount of variability is better. The change reflects the difference in values between the pre- and post-training sessions. The discharge rate variability will change by percent.
Change in Blood-oxygen-level-dependent(BOLD) Activity of Motor Cortex | Change from Baseline to 1 month
  Results of blood-oxygen-level-dependent contrast imaging as analyzed from functional Magnetic Resonance Imaging(fMRI). More colors indicates more excitement of the motor cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Christou, PhD, Principal Investigator — University of Florida; David Vaillancourt, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manto MU. The wide spectrum of spinocerebellar ataxias (SCAs). Cerebellum. 2005;4(1):2-6. doi: 10.1080/14734220510007914. PMID 15895552
- [Background] Manto M. Mechanisms of human cerebellar dysmetria: experimental evidence and current conceptual bases. J Neuroeng Rehabil. 2009 Apr 13;6:10. doi: 10.1186/1743-0003-6-10. PMID 19364396
- [Background] Solodkin A, Gomez CM. Spinocerebellar ataxia type 6. Handb Clin Neurol. 2012;103:461-73. doi: 10.1016/B978-0-444-51892-7.00029-2. PMID 21827907
- [Background] Schmitz-Hubsch T, Tezenas du Montcel S, Baliko L, Boesch S, Bonato S, Fancellu R, Giunti P, Globas C, Kang JS, Kremer B, Mariotti C, Melegh B, Rakowicz M, Rola R, Romano S, Schols L, Szymanski S, van de Warrenburg BP, Zdzienicka E, Durr A, Klockgether T. Reliability and validity of the International Cooperative Ataxia Rating Scale: a study in 156 spinocerebellar ataxia patients. Mov Disord. 2006 May;21(5):699-704. doi: 10.1002/mds.20781. PMID 16450347
- [Background] Kawaguchi Y, Okamoto T, Taniwaki M, Aizawa M, Inoue M, Katayama S, Kawakami H, Nakamura S, Nishimura M, Akiguchi I, et al. CAG expansions in a novel gene for Machado-Joseph disease at chromosome 14q32.1. Nat Genet. 1994 Nov;8(3):221-8. doi: 10.1038/ng1194-221. PMID 7874163
- [Background] Reetz K, Costa AS, Mirzazade S, Lehmann A, Juzek A, Rakowicz M, Boguslawska R, Schols L, Linnemann C, Mariotti C, Grisoli M, Durr A, van de Warrenburg BP, Timmann D, Pandolfo M, Bauer P, Jacobi H, Hauser TK, Klockgether T, Schulz JB; axia Study Group Investigators. Genotype-specific patterns of atrophy progression are more sensitive than clinical decline in SCA1, SCA3 and SCA6. Brain. 2013 Mar;136(Pt 3):905-17. doi: 10.1093/brain/aws369. Epub 2013 Feb 18. PMID 23423669
- [Background] Pasternak O, Shenton ME, Westin CF. Estimation of extracellular volume from regularized multi-shell diffusion MRI. Med Image Comput Comput Assist Interv. 2012;15(Pt 2):305-12. doi: 10.1007/978-3-642-33418-4_38. PMID 23286062
- [Background] Pasternak O, Sochen N, Gur Y, Intrator N, Assaf Y. Free water elimination and mapping from diffusion MRI. Magn Reson Med. 2009 Sep;62(3):717-30. doi: 10.1002/mrm.22055. PMID 19623619
- [Background] De Luca CJ, Adam A, Wotiz R, Gilmore LD, Nawab SH. Decomposition of surface EMG signals. J Neurophysiol. 2006 Sep;96(3):1646-57. doi: 10.1152/jn.00009.2006. PMID 16899649
- [Background] Morton SM, Bastian AJ. Cerebellar control of balance and locomotion. Neuroscientist. 2004 Jun;10(3):247-59. doi: 10.1177/1073858404263517. PMID 15155063
- [Background] Haines DE, Manto MU. Clinical symptoms of cerebellar disease and their interpretation. Cerebellum. 2007;6(4):360-74. doi: 10.1080/14734220701798199. No abstract available. PMID 18041661
- [Background] Keller JL, Bastian AJ. A home balance exercise program improves walking in people with cerebellar ataxia. Neurorehabil Neural Repair. 2014 Oct;28(8):770-8. doi: 10.1177/1545968314522350. Epub 2014 Feb 13. PMID 24526707